CLINICAL TRIAL: NCT05494710
Title: Bleomycin Electrosclerotherapy Treatment of Vascular Malformations: A Feasibility Study
Acronym: BEST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: South Tees Hospitals NHS Foundation Trust (Other)
Collaborators: Teesside University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 248206
Record Dates: First submitted 2022-01-26; First posted 2022-08-10 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Vascular Malformations
MeSH Terms: conditions — Vascular Malformations

STUDY DESIGN:
Intervention Model Description: single group of patients receiving same treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bleomycin electrosclerotherapy treatment (Experimental): Bleomycin electrosclerotherapy treatment administered. The combination of Bleomycin and electroporation of the treated area is called electrochemotherapy (ECT).
  Interventions: Other: Bleomycin electrosclerotherapy treatment

INTERVENTIONS:
Other: Bleomycin electrosclerotherapy treatment — The combination of Bleomycin and electroporation of the treated area which is called electrochemotherapy (ECT).

SUMMARY:
The aim of the BEST study is to examine the feasibility of assessing patient and clinician reported outcome of a single electrosclerotherapy treatment of vascular malformations.

* Sclerotherapy = injection of Bleomycin into vascular birthmarks to seal off abnormal vascular channels
* Electroporation = application of an electric field to vessels treated with a handheld needle electrode
* Electrosclerotherapy = a combination of Bleomycin sclerotherapy and electroporation

ELIGIBILITY:
Inclusion Criteria:

* New patients presenting with a vascular malformation suitable for Bleomycin sclerotherapy treatment
* Existing patients presenting with a poor response to treatment, performed more than 6 months ago
* Placement of a needle electrode into the vascular malformation is technically possible
* Evaluation of response to treatment is possible on photo documentation
* Patients agreeing to participate in the study
* The ability to understand written and spoken English

Exclusion Criteria:

* Patients not agreeing to participate in the study
* Pregnancy
* Breastfeeding
* Previous high systemic Bleomycin exposure (more than 3000 IU)
* Patients unable to provide written, informed consent
* Patients in which needle electrode placement is not possible
* Response to treatment not evaluable by photo documentation
* Patients unable to speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Quality of life questionnaire scores between baseline and 6-8 weeks of treatment | 8 weeks
  Patient reported quality of life after a single electrosclerotherapy treatment of vascular malformations - change in scores measured using Birthmark Quality of Life questionnaire (8 items measured on 5 point scale)
Clinician assessment tool of treatment response | 8 weeks
  Clinician assessment of treatment response following electrosclerotherapy treatment using clinical assessment tool - change in scores measured

SECONDARY OUTCOMES:
To collect documented side effects following electrosclerotherapy treatment. | 2 years
  To collect documented side effects following electrosclerotherapy treatment using diary

CONTACTS AND LOCATIONS:
Locations (1):
- South Tees Hospitals NHS Foundation Trust, Middlesbrough, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided